CLINICAL TRIAL: NCT01721577
Title: Phase I/II Clinical Trial of the Safety, Tolerability, and Anti-tumor Efficacy of the IGF-1R Inhibitor, AXL1717 (Picropodophyllin), in the Treatment of Recurrent Malignant Astrocytomas
Brief Title: Phase I/II Trial of AXL1717 in the Treatment of Recurrent Malignant Astrocytomas
Acronym: AXL1717
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator went to another institution.
Sponsor: Rush University Medical Center (Other)
Collaborators: Axelar AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11090804; VABC; GCR (Other Grant/Funding Number: Voices Against Brain Cancer; Gateway for Cancer Research)
Record Dates: First submitted 2012-10-29; First posted 2012-11-05 (Estimated); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Anaplastic Ependymoma
Keywords: glioblastoma; gliosarcoma; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic oligoastrocytoma; AXL1717; IGF-1 receptor inhibitor; picropodophyllin
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Ependymoma | interventions — picropodophyllin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1: AXL1717, 300mg (Experimental): In the first phase, 10-20 patients will be enrolled and treated with 300mg (original range of starting dose was 300-520mg) BID of AXL1717 for 28 days. The primary endpoint of the first phase is to determine the recommended Phase 2 dose (RP2D) of AXL1717 and to assess the safety and toxicity of AXL1717. The study has a 3+3 design and the first cohort will be treated with 300 mg AXL1717 BID for 28 days repeated in up to 5 cycles. The highest dose level without DLT or with maximally one DLT out of 6 patients will be the RP2D. Non-progressing patients may be treated for a total of five 28-day cycles (24 weeks).
  Interventions: Drug: AXL1717

INTERVENTIONS:
Drug: AXL1717 — IGF-1 receptor inhibitor
  Other Names: picropodophyllin

SUMMARY:
This is a single-center, open-label, non-randomized, Phase I/IIa study to investigate the safety, tolerability, and antitumor efficacy of AXL1717 (picropodophyllin as active agent formulated in an oral suspension; PPP) in patients with recurrent malignant astrocytomas (glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, and anaplastic ependymoma). Patients will be treated for up to 5 cycles. A treatment cycle is defined as 28 days+7 days rest (28+7 days during cycle 1 to 4, and 28 days during cycle 5). The following cycle will not be started until the treatment continuation criteria are fulfilled. Concomitant supportive therapies will be allowed.

DETAILED DESCRIPTION:
AXL1717, as a ready-to-use suspension of picropodophyllin for oral administration, will be distributed in bottles for single use at a concentration of 25 mg/mL. Fixed doses will be used, i.e. there are no adjustments for weight or body surface. There will be no randomization or blinding in the study.

The trial will be divided in two phases. In the first phase, 10-20 patients will be enrolled and treated with 300-520 mg BID of AXL1717 for 28 days. The primary endpoint of the first phase is to determine the recommended Phase 2 dose (RP2D) of AXL1717 in patients with recurrent or progressive glioblastoma and to assess the safety and toxicity of AXL1717 in this patient population. The study has a 3+3 design and the first cohort will be treated with 400 mg AXL1717 BID for 28 days repeated in up to 5 cycles. If dose-limiting toxicity (DLT) such as neutropenia occurs, dosing will be interrupted and the individual patient will, following normalization, be restarted on the same or a lower dose level according to standardized procedure. If two or three of the first 3 patients on a specific dose level experience a DLT during the first 28 days of treatment with AXL1717, the following patients will be treated with a lower dose level. If one DLT occurs during the first 28 days of dosing in the first 3 three patients another 3 patients will be treated with the same dose level. If 2 of the 6 patients display DLT, the next patients will be treated with a lower dose level. The highest dose level without DLT or with maximally one DLT out of 6 patients will be the RPTD. All assessments with respect to dose adjustments for subsequent cohorts will be done during the first 28 days of treatment. Non-progressing patients may be treated for a total of five 28-day cycles (24 weeks).

In the second phase, 12 patients will be enrolled and treated with the identified RP2D of AXL1717 for 28 days repeated in five cycles. The primary endpoints of phase II is to assess the proportion of patients who are progression-free at 24 weeks and to assess safety, tolerability, and adverse event profile of AXL1717.

ELIGIBILITY:
Inclusion criteria

1. Be informed of the nature of the study and have provided written informed consent
2. At least 18 years of age
3. ECOG performance of 0, 1, or 2, or KPS (Karnofsky performance status) ≥ 60.
4. Pathological verification of a WHO grade 4 astrocytoma (glioblastoma or gliosarcoma), or WHO Grade 3 anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, or anaplastic ependymoma.
5. Documented recurrent glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, or anaplastic ependymoma after at least one failed treatment of chemotherapy and radiation
6. Expected survival of at least 3 months
7. At least 2-weeks from cytoreductive surgery, if performed, 4-weeks from bevacizumab or other chemotherapy (6-weeks if prior chemotherapy was nitrosourea) and 12-weeks from completion of radiotherapy.
8. Ability to undergo MRI scanning without and with imaging dye on a periodic basis as defined in the protocol
9. Preserved major organ functions, i.e: Blood leukocyte count ≥ 3.0 x 109/L Blood absolute neutrophil count ≥ 1.5 x 109/L Blood platelet count ≥ 100 x109/L Blood hemoglobin ≥ 100 g/L (transfusions are allowed) Plasma total bilirubin level ≤ 1.5 times the upper institutional limit (ULN) of the ‖normal‖ (i.e. reference) range Plasma AST (aspartate aminotransferase) or ALT ≤ 2.5 times upper institutional limit (ULN) of the ‖normal‖ range Plasma creatinine ≤ 1.5 times upper institutional limit (ULN) of the ‖normal‖ range 12-lead ECG with normal tracings; or changes that are not clinically significant and do not require medical intervention, and QTc < 500 ms At least seven (7) days off of medications which inhibit or induce CYP2C9 or CYP3A4 before first study treatment day

Exclusion criteria

1. Any or other major recent or ongoing disease that, according to the Investigator, poses an unacceptable risk to the patient
2. Grade 3 or higher constipation within the past 28 days or grade 2 constipation within the past 14 days before randomization. (Patients with grade 2 constipation within the past 14 days could be re-screened if constipation decreases to ≤ grade 1 with optimal management of constipation.)
3. Coexisting uncontrolled medical condition.
4. Hepatitis B or Hepatitis C, or HIV infection requiring anti-retroviral therapy
5. Active malignancy other than basal cell skin cancer
6. Other active malignancy during the previous 3 years
7. Major surgical procedure within 4 weeks
8. Prior stereotactic or gamma knife radiosurgery or proton radiation, unless unequivocal progression by functional neuro-imaging (PET, dynamic MRI, MRS, SPECT) or by re-operation with documented histologic confirmation of recurrence.
9. Prior anti-tumor therapy, as follows: at least 12-weeks from radiation therapy; at least 4-weeks from prior treatment with temozolomide or bevacizumab, 6-weeks from BCNU or CCNU.
10. Women of child bearing potential (WOCBP) who do not consent to using acceptable methods of birth control (oral contraceptives, IUD). For purposes of this study, WOCBP include any female who has experienced menarche, who has not undergone tubal ligation, and who is not postmenopausal.
11. Medically uncontrolled Type 1 or Type 2 diabetes mellitus
12. Pregnancy or lactation
13. Current participation in any other investigational clinical trial within 4-weeks.
14. Eastern Cooperative Oncology Group (ECOG) performance status > 2 after optimization of medications (See Appendix 4) or KPS < 60
15. Anticipated Life expectancy less than 3 months
16. Contraindications to the investigational product or known or suspected hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Aiken, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Andrews DW, Resnicoff M, Flanders AE, Kenyon L, Curtis M, Merli G, Baserga R, Iliakis G, Aiken RD. Results of a pilot study involving the use of an antisense oligodeoxynucleotide directed against the insulin-like growth factor type I receptor in malignant astrocytomas. J Clin Oncol. 2001 Apr 15;19(8):2189-200. doi: 10.1200/JCO.2001.19.8.2189. PMID 11304771
- [Background] Girnita A, Girnita L, del Prete F, Bartolazzi A, Larsson O, Axelson M. Cyclolignans as inhibitors of the insulin-like growth factor-1 receptor and malignant cell growth. Cancer Res. 2004 Jan 1;64(1):236-42. doi: 10.1158/0008-5472.can-03-2522. PMID 14729630
- [Background] Ekman S, Frodin JE, Harmenberg J, Bergman A, Hedlund A, Dahg P, Alvfors C, Stahl B, Bergstrom S, Bergqvist M. Clinical Phase I study with an Insulin-like Growth Factor-1 receptor inhibitor: experiences in patients with squamous non-small cell lung carcinoma. Acta Oncol. 2011 Apr;50(3):441-7. doi: 10.3109/0284186X.2010.499370. Epub 2010 Aug 11. PMID 20698809
- [Background] Yin S, Girnita A, Stromberg T, Khan Z, Andersson S, Zheng H, Ericsson C, Axelson M, Nister M, Larsson O, Ekstrom TJ, Girnita L. Targeting the insulin-like growth factor-1 receptor by picropodophyllin as a treatment option for glioblastoma. Neuro Oncol. 2010 Jan;12(1):19-27. doi: 10.1093/neuonc/nop008. Epub 2009 Oct 20. PMID 20150364

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was excluded from the study after screening but before treatment and is not considered in this analysis.
Groups:
- AXL1717 400mg BID: Started on 400mg BID
- AXL1717 300mg BID: Started on 300mg BID
Period: Overall Study
Arm/Group | AXL1717 400mg BID | AXL1717 300mg BID
Started | 2 | 7
Completed | 0 | 4
Not Completed | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Death | 1 | 0
Not completed — Dose Escalation to 400mg BID | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- AXL1717, 400mg Initial Dose: Subjects who started and completed the study on 400mg BID
- AXL1717, 300mg Initial Dose: Subjects who started the study on 300mg BID. one subject was escalated to 400mg BID and 2 subjects were de-escalated to 215mg BID
- Total: Total of all reporting groups
Arm/Group | AXL1717, 400mg Initial Dose | AXL1717, 300mg Initial Dose | Total
Number analyzed (Participants) | 2 | 7 | 9
Age, Continuous [Mean (Full Range); unit: Years] | 58 [57 to 59] | 56.2 [37 to 69] | 56.6 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Determine Recommended Phase II Dose
Description: To determine the recommended phase II dose (RPTD) of AXL1717 in recurrent malignant astrocytomas defined as the highest dose level without DLT (Dose Limiting Toxicity) or with maximally one DLT out of 6 patients will be the RPTD.
Time Frame: 8 months
Measure: Number; unit: MG
Groups:
- All Study Participants: All study participants who received different doses of the same formulation of AXL1717.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
MG | NA — No dose in the trial met this criteria for establishing a RPTD.

2. Primary Outcome: Phase II - To Determine if AXL1717 Has Any Antitumor Effect
Description: To determine if AXL1717 has any antitumor effect as a single agent treatment in recurrent malignant astrocytomas by evaluating PFS at 24 weeks
Time Frame: 24 Weeks
Population: Phase II of this study was never initiated and so no data was collected or analyzed for this endpoint.
Groups:
- Phase II Subject Group: This group was never established as Phase I of the study was never completed and thus Phase II was never initiated.
Arm/Group | Phase II Subject Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase I - To Identify the Maximum Tolerable Dose
Description: To identify the Maximum Tolerated Dose (MTD) of AXL1717 in the Phase I subject population. MTD is the highest dose of AXL1717 with the lowest average per subject cases of DLT.
Time Frame: 8 Months
Measure: Number; unit: MG
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
MG | 300

4. Secondary Outcome: Phase I - Molecular Markers of Optimum Response
Description: To assess potential molecular markers that might predict optimum response sub-population groups
Time Frame: 8 months
Population: the data for this outcome measure was not collected and/or analyzed. There is no data to report.
Groups:
- AXL1717: All subject who participated in the study and received at least one cycle of treatment.
Arm/Group | AXL1717
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase I - Molecular Markers of IGF (Insulin Like Growth Factor)-1R Pathway
Description: To evaluate surrogate molecular markers of IGF-1R pathway activation/inhibition after treatment with AXL1717 in patients with malignant astrocytomas
Time Frame: 8 months
Population: None of the secondary outcome measures were collected or analyzed as this study was conducted using the oral suspension of AXL1717 and there is a new formulation of AXL1717 in development (capsule). Decision was made to abandon other analysis or data collections in regards to secondary outcomes.
Groups:
- AXL1717, 400mg Initial Does: first 2 subjects were started on 400mg BID initial dose.
- AXL1717, 300mg Initial Does: Subjects who were started on 300mg BID
Arm/Group | AXL1717, 400mg Initial Does | AXL1717, 300mg Initial Does
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase II - Time-To-Progression (TTP) and Overall Survival (OS)
Description: To determine time-to-progression (TTP) and overall survival (OS) of patients treated with AXL1717. Only overall survival for subjects is prolonged stable disease was analyzed.
Time Frame: 4 months
Population: Phase II of this study was never initiated and so no data was collected or analyzed for this endpoint.
Groups:
- Phase II Study Population: This group was never established as Phase I of the study was never completed and thus Phase II was never initiated.
Arm/Group | Phase II Study Population
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase II - Overall Response Rate
Description: To assess overall response rate (ORR) in recurrent malignant astrocytomas after treatment with AXL1717
Time Frame: 4 months
Population: Phase II of the study was never initiated. No data was gathered or analyzed.
Arm/Group | Phase II Study Population
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase II - Identify Evidence of Response on Imaging
Description: To identify surrogate imaging evidence of response on MRI sequences (especially T2- FLAIR, DWI, Perfusion MRI and multi-voxel MRS).
Time Frame: 8 Months
Population: Phase II of the study was never initiated.
Arm/Group | Phase II Subject Group
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Exploratory Endpoint - Determine Antitumor Effect
Description: To assess the ability of AXL1717 to inhibit tumor proliferation as assessed by blood IGFBP-1 through IGFBP-7, growth hormone (GH) levels, C-peptide, IGF-1 (free and total), and IGF-2 levels, insulin, and analysis of tumor tissue of patients treated with AXL1717 for 5 days before surgical re-operation by examining for the IGF-1R signal transduction pathway in the resected brain tumor tissue, and correlate with outcome.
Time Frame: 4 months
Population: Phase II portion of this study was not initiated as the phase 1 piece was not completed fully. This endpoint was not explored and data was not collected or analyzed
Arm/Group | AXL1717, 400mg Initial Dose | AXL1717, 300mg Initial Dose
Number analyzed (Participants) | 0 | 0

10. Post Hoc Outcome: Phase I Subjects - Imaging Evidence of Response.
Description: Number of Participants with Imaging Evidence of Response on MRI (magnetic resonance imaging)sequences by RANO criteria (with additional special attention to T2-FLAIR, DWI (diffusion-weighted imaging), perfusion MRI and multi-voxel MRS (magnetic resonance spectroscopy) sequences).
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- AXL1717, 400mg Initial Dose: Subjects who were started on 400mg initial dose
- AXL1717, 300mg Initial Dose: Subjects who were started on 300mg initial dose
Arm/Group | AXL1717, 400mg Initial Dose | AXL1717, 300mg Initial Dose
Number analyzed (Participants) | 2 | 7
Participants | 0 | 5

ADVERSE EVENTS:
Time Frame: information was collected for each subject while on study (~some were up to 1 year)
Groups:
- 400mg BID: Subjects on 400mg BID of AXL1717
- 300mg BID: Subjects on 300mg BID of AXL1717
- 215mg BID: Subjects on 215mg BID of AXL1717
Arm/Group | 400mg BID | 300mg BID | 215mg BID
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/7 | 1/2
Other Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400mg BID (N=3) | 300mg BID (N=7) | 215mg BID (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400mg BID (N=3) | 300mg BID (N=7) | 215mg BID (N=2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesias (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
I am not privvy to all the agreements that exist. But the original PI left the institution where this study was conducted, and he left with a separation agreement in place. I (Crista Brawley) am named in that agreement. Please direct questions to Dr. Robert Aiken.